CLINICAL TRIAL: NCT05005364
Title: Prospective Evaluation of the Clinical Profile and Treatment Outcomes of Proximal Humerus Fractures.
Acronym: SPHEER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Bryan Tan, Associate Consultant, Tan Tock Seng Hospital
Other Study IDs: 2016/01241
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Proximal Humerus Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With an ageing population, fragility fractures secondary to osteoporosis are on a increasing trend. Proximal humerus fractures are common fractures which account for a significant proportion of these fragility fractures. They significantly affect patients function and independence particularly in the elderly.

Currently, treatment options range from conservative treatment with an arm sling to fixation either with plates or intramedullary devices to arthroplasty ranging from a hemiarthroplasty to the latest reverse shoulder arthroplasty. While is there has been a global trend towards surgical treatment for such fractures, there is significant controversy regarding the best treatment with many studies reporting disappointing functional outcomes including residual shoulder pain, limitation in shoulder motion and decreased quality of life regardless of treatment option selected.

In this day and age where healthcare cost is a big concern both at the individual patient level but at a government level as well, evaluating the cost effectiveness of treatment becomes essential as well. Currently in Singapore, there have been a significant trend of an increased use of surgical treatment of proximal humerus fractures however we have very little data in our local context not only to evaluate the clinical effectiveness but also the cost effectiveness of surgical treatment in comparison to conservative treatment.

The primary aim of the study is

1. To understand the epidemiology and prognostic factors for proximal humerus fractures

   * Incidence
   * Health service utilization
   * clinical and functional outcomes
2. To estimate the relative cost-effectiveness of surgical vs non-surgical treatment pathways for managing patients with proximal humerus fractures.

We hypothesize that surgical fixation of the proximal humerus is both clinically and cost effective

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years old and above
2. Radiologically confirmed proximal humerus fracture
3. Within 3 weeks of their injury

Exclusion Criteria:

1. Open fracture
2. Mentally incompetent patients
3. Co-morbidities precluding anaesthesia
4. Severe soft tissue compromise
5. Neurovascular compromise
6. Pathological fracture other than osteoporosis
7. Surgery delayed > 3 weeks
8. Pregnancy

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with proximal humerus fracture going for surgical or conservative treatment option
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Constant Shoulder Score - change over 6 weeks, 3, 6, 12 months | Assessed at baseline, 6 weeks, 3 months, 6 months, 12 months
  To evaluate the clinical outcomes over time by comparing the change in constant shoulder score over a period of 1 year. The Constant Shoulder Score is used to assess the level of pain and the patient's ability to carry out normal daily activities.
  Constant score of the unaffected shoulder was also assessed at baseline to compare the function between the two shoulders.
Oxford Shoulder Score - change over 6 weeks, 3, 6, 12 months | Assessed at baseline, 6 weeks, 3 months, 6 months, 12 months
  A 12-item patient-report questionnaire developed to evaluate the outcome of shoulder surgery, excluding surgery for instability. The OSS contains two subscales, pain and activities of daily living. Each responses is of a 0-4 scoring format with a higher score representing better function. Hence, the highest possible total score is 48 and a higher score represents a better outcome.
QuickDASH scoring - change over 6 weeks, 3, 6, 12 months | Assessed at baseline, 6 weeks, 3 months, 6 months, 12 months
  This score is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
EQ5D-5L - change over 6 weeks, 3, 6, 12 months | Assessed at baseline, 6 weeks, 3 months, 6 months, 12 months
  EuroQol-5 Dimensions (EQ-5D) consists of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
Costing questionnaire | Assessed at 6 weeks, 3 months, 4.5 months, 6 months
  Questionnaire measuring the direct and indirect costs

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Tan, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore